CLINICAL TRIAL: NCT03681938
Title: Indication to Transplant Patients With High Risk B Cells Lymphoma in Metabolic Complete Remission After 2 Cycles of Chemotherapy ?
Brief Title: Indication to Transplant Patients With High Risk B Cells Lymphoma in Metabolic Complete Remission?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: ALERT-IPC 2017-015
Record Dates: First submitted 2017-10-26; First posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Transplantation, Autologous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intensification treatment: Autograft
  Interventions: Procedure: Autograft
- Standard chemotherapy (without autograft)

INTERVENTIONS:
Procedure: Autograft — Autograft
  Groups: Intensification treatment: Autograft

SUMMARY:
The autograft of patients with prognostically unfavourable B-cells lymphoma cells in first remission remains controversial, in particular since the association of Rituximab with chemotherapy. Even though many randomized and non-randomized studies have been conducted, their is still no standard procedure . Recently, the use of early TEP (positron emission topography) answer, after 2 in 3 cures of chemotherapy allowed to select the poor-responder patients who remain candidate to autograft in front-line. Nevertheless, in good-responder patients, the benefits of an intensification therapy ins term of long-lasting disease control remains discussion.

This institutional retrospective study aims at comparing the outcome of early metabolic responder patients who received an intensification treatment to those who received a standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with High Risk Big B Cells Lymphoma
* Age > 18 years

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With High Risk Big B Cells Lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2019-07-28 (Estimated); Study Completion 2019-07-28 (Estimated)

PRIMARY OUTCOMES:
Compare the survival without progress of transplanted patients versus not transplanted patients | From the date of complete remission post C2 of chemotherapy up to 120 months
  Medical follow up

SECONDARY OUTCOMES:
Cumulative Relapse Incidence | From the date of complete remission post C2 of chemotherapy up to 120 months
  Medical follow up
Overall survival | From the date of complete remission post C2 of chemotherapy up to 120 months
  Medical follow up

CONTACTS AND LOCATIONS:
Overall Officials: BOUABDALLAH Réda, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Institut paoli-calmettes — http://www.institutpaolicalmettes.fr